CLINICAL TRIAL: NCT00564369
Title: CDC HIV Testing Guidelines: Unresolved Ethical Concerns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other)
Responsible Party: Roland C. Merchant, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 106879-42-RGAT; 106879-42-RGAT
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections
Keywords: HIV testing; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 2006 CDC recommendations
  Interventions: Other: CDC HIV testing recommendations
- 2 (Active Comparator): Prior CDC recommendations
  Interventions: Other: CDC HIV testing recommendations

INTERVENTIONS:
Other: CDC HIV testing recommendations — Current vs. prior CDC recommendations

SUMMARY:
Advocacy groups have voiced concerns about the ethics of some of tenets of the CDC's new HIV testing recommendations for the healthcare setting. Three concerns are paramount: (1) the opt-out approach to HIV testing can potentially be coercive and not truly voluntary; (2) by replacing informed consent with general consent for medical care, test participants might not know or be adequately informed of the benefits and consequences of testing; and (3) eliminating HIV prevention counseling from the HIV testing process presumes that test participants are aware of how to prevent an HIV infection, which might not be correct. This study involves conducting interviews of HIV advocates who are raising these concerns, surveying outpatient and emergency department clinical providers about their beliefs and opinions regarding the tenets of the new guidelines, and then conducting a multi-center, randomized, controlled trial in which the ethical concerns of opt-out vs. opt-in testing are directly compared. We will conduct a multi-center, randomized, controlled, trial whereby patients will be surveyed on their perspectives and perceptions regarding opt-out or opt-in rapid HIV testing. We will survey the participants regarding their perception of coercion, their understanding of the elements contained in the informed consent process, their HIV risk factors, and their knowledge of HIV prevention. We will evaluate whether or not the CDC-recommended approaches regarding opt-out testing, consent, and decoupling of prevention counseling are supported. If there are no differences regarding these ethical concerns between testing approaches, then the opt-out approach would be considered not to be inferior to the opt-in approach.

ELIGIBILITY:
Inclusion Criteria:

* 18-64-year-old patients in the outpatient family practice and medical clinics and emergency departments of Memorial Hospital, Miriam Hospital, and Rhode Island Hospital who speak English or Spanish and are not HIV infected

Exclusion Criteria:

* HIV infection
* Inability to speak English or Spanish
* A physical, psychiatric, or mental disability that prevents participation in the study
* Involvement in an HIV vaccine study
* Prisoner

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Perceptions among patients and providers regarding the concerns about the 2006 CDC HIV testing recommendations | Immediate

SECONDARY OUTCOMES:
Comparison/contrast of patient and provider perspectives on concerns raised about the 2006 CDC HIV testing recommendations | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Roland C Merchant, MD, MPH, ScD, Principal Investigator — Rhode Island Hospital
Locations (3):
- United States (3):
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island